CLINICAL TRIAL: NCT07136779
Title: PHASE 1/2A OPEN-LABEL CLINICAL TRIAL EVALUATING VBC101, AN EGFR AND CMET TARGETED BI-SPECIFIC ANTIBODY DRUG CONJUGATE, IN PARTICIPANTS WITH ADVANCED SOLID TUMOR MALIGNANCIES
Brief Title: First-in-Human Trial of VBC101 in Participants With Advanced Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VelaVigo Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBC101-01-01
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Participants With Advanced Solid Tumor Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 (Dose Escalation and Backfill)，Phase 2（Dose optimization and Cohort Expansion） (Experimental)
  Interventions: Drug: VBC101

INTERVENTIONS:
Drug: VBC101 — VBC101

SUMMARY:
This is a multicenter, open-label, multiple-dose, FIH Phase 1/2a trial. The Phase 1 portion adopts an accelerated titration for the first dose level, followed by BOIN design to identify the MTD and/or RP2D with potential backfill cohorts. The Phase 2a portion consists of dose optimization followed by cohort expansion to confirm safety and tolerability and to further evaluate the efficacy of the selected RP2D in selected solid tumor malignancies for VBC101.

ELIGIBILITY:
Inclusion Criteria:

* A participant must meet all of the following inclusion criteria to be eligible to participate in this trial:
* 1. The participant or the participant's legally acceptable representative is willing and able to provide a written ICF before initiating any trial procedure.
* 2. Histologically or cytologically confirmed unresectable advanced/metastatic solid tumor that has relapsed or progressed on or after standard systemic treatments, or is intolerable with standard treatment, or for which no standard treatment is available
* 3. At least one measurable lesion as assessed by the investigator according to RECIST v1.1criteria
* 4. Male or female adults (defined as ≥ 18 years of age)
* 5. ECOG performance status 0-1
* 6. Has LVEF ≥ 50% by either ECHO or MUGA within 28 days before enrollment.
* 7. Life expectancy greater than 12 weeks
* 8. Archived tumor tissue sample available or able to undergo a fresh biopsy collection.
* 9. Adequate organ and bone marrow function
* 10. Participants must meet the minimum washout period requirements before the first dose of investigational drug

Exclusion Criteria:

1. Any unresolved toxicity of Grade ≥2 from previous anti-cancer treatment, except for alopecia, neuropathy, or skin pigmentation changes. Participants with chronic but stable Grade 2 toxicities may be allowed to enroll after agreement between the study investigator and the Sponsor's Medical Monitor.

* 2. Known or suspected brain metastases, or spinal cord compression, unless the condition has been treated, asymptomatic, and has been stable without requiring escalating doses of corticosteroids (equivalent to ≤10 mg/day prednisone) or anti-convulsant medications for at least four weeks prior for the first dose of investigational drug.
* 3. Prior treatment with an ADC targeting EGFR and/or cMet (including VBC101)
* 4. Prior treatment with any ADC carrying a TOP1i payload (including prior VBC101).
* 5. Has a medical history of interstitial lung diseases (e.g., non-infectious interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or current interstitial lung diseases or who are suspected to have these diseases by imaging at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) as defined in the protocol | (DLT)From time of first dose of VBC101 to end of DLT period (approximately 21 days)
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Incidence of Serious Adverse Events | From time of Informed Consent to 30 days post last dose of VBC101
  Number of patients with serious adverse events by system organ class and preferred term
Incidence of Adverse Events (AEs) | From time of Informed Consent to 30 days post last dose of VBC101
  Number of patients with adverse events by system organ class and preferred term

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose of VBC101 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The percentage or number of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST v1.1)
Duration of Response (DoR) | From date of first dose of VBC101 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The time from date of first response until date of disease progression or last evaluable assessment (RECIST v1.1) in the absence of progression
Disease Control Rate (DCR) at 12 weeks | From date of first dose of VBC101 up until progression, or the last evaluable assessment in the absence of progression (for each patient this is expected to be measured at 12 weeks)
  The percentage of patients with confirmed CR or PR or having SD maintained (RECIST v1.1) for >=11 weeks from first dose
Progression free Survival (PFS) | From date of first dose of VBC101 up until date of progression or death due to any cause (approximately 2 years)
  The time from first dose until RECIST 1.1 defined disease progression or death due to any cause
Overall Survival (OS) | From date of first dose of VBC101 up until the date of death due to any cause (approximately 2 years)
  The time from the date of the first dose of study treatment until death due to any cause.
Pharmacokinetics of VBC101: Plasma PK concentrations | From date of first dose of VBC101 up until 30 days post last dose
  Measurement of plasma concentrations of VBC101, total antibody and total unconjugated warhead
Pharmacokinetics of VBC101: Area under the concentration time curve (AUC) | From date of first dose of VBC101 up until 30 days post last dose
  Measurement of PK parameters: Area under the concentration time curve (AUC)
Pharmacokinetics of VBC101: Maximum plasma concentration of the study drug (C-max) | From date of first dose of VBC101 up until 30 days post last dose
  Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max)
Pharmacokinetics of VBC101: Time to maximum plasma concentration of the study drug (T-max) | From date of first dose of VBC101 up until 30 days post last dose
  Measurement of PK parameters: Time to maximum observed plasma concentration of the study drug (T-max)
Pharmacokinetics of VBC101: Half-life | From date of first dose of VBC101 up until 30 days post last dose
  Measurement of PK parameters: Terminal elimination half-life (t 1/2)
Immunogenicity of VBC101: Anti-Drug Antibodies (ADA) | From date of first dose of VBC101 up until 30 days post last dose
  Evaluating the number and percentage of patients who develop Anti-drug antibody (ADA) during treatment

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Start Midwest, Grand Rapids, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - START Mountain Region, LLC., West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided